CLINICAL TRIAL: NCT03614195
Title: Immediate and Retained Effects of Three Types of Dual-task Interventions on Dual-task Walking Performance of Stroke Patients: Psychometric Study and Randomized Controlled Trial
Brief Title: Effects of Three Types of Dual-task Interventions on Dual-task Walking Performance of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Li-Ling Chuang, Assistant Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201701988A3
Record Dates: First submitted 2018-07-31; First posted 2018-08-03 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MCDTT (Experimental): The MCDTT group will receive dual-task interventions at progressively increasing task difficulty 3 times a week for 4 weeks.
  Interventions: Device: MCDTT
- MDTT (Active Comparator): The MDTT group will receive dual-task interventions at progressively increasing task difficulty 3 times a week for 4 weeks.
  Interventions: Device: MDTT
- CDTT (Active Comparator): The CDTT group will receive dual-task interventions at progressively increasing task difficulty 3 times a week for 4 weeks.
  Interventions: Device: CDTT

INTERVENTIONS:
Device: MCDTT — The MCDTT group will undertake sitting to standing, standing balance, and treadmill walking training while concurrently perform motor and cognitive tasks.
  Arms: MCDTT
Device: MDTT — The MDTT group will train the same set of sitting to standing, standing balance, and walking activities as the MCDTT group while simultaneously performing only motor task.
  Arms: MDTT
Device: CDTT — The CDTT group will train the same set of sitting to standing, standing balance, and walking activities as the MCDTT group while simultaneously performing only cognitive task.
  Arms: CDTT

SUMMARY:
The objective of this study is to investigate psychometric properties of dual-task walking assessments and compare effects of three types of dual-task balance interventions on dual-task walking for stroke patients.

DETAILED DESCRIPTION:
English Synopsis

I. Title of Study:

Immediate and retained effects of three types of dual-task interventions on dual-task walking performance of stroke patients: psychometric study and randomized controlled trial

II. Study Objectives:

The objective of this study is to investigate psychometric properties of dual-task walking assessments and compare effects of three types of dual-task balance interventions on dual-task walking for stroke patients. Specifically, we will investigate psychometric properties (i.e. reliability, validity, and responsiveness) of dual-task walking assessments with various levels of difficulty for stroke individuals (Aim 1). The second aim of this study is to compare the immediate and retained effects of combined motor and cognitive dual-task training (MCDTT), motor dual-task training (MDTT), and cognitive dual-task training (CDTT) on dual-task gait and cognitive performance after stroke (Aim 2). The third aim of this study is to elucidate the changed CMI pattern of stroke patients after dual-task interventions (Aim 3).

III. Study Design A metric analysis and comparative efficacy research will be conducted at medical center(s). Sixty ambulatory stroke patients will receive dual-task walking assessments twice at pretreatment with a 1-week interval for test-retest assessment and investigation of the reliability and validity of outcome measures. The primary outcome measure of the six dual-task walking assessments will include two types of walking conditions (walking at preferred speed and fast speed) and simultaneously perform three cognitive tasks (Serial Three Subtractions, Stroop, and Auditory Stroop tasks). These three cognitive tasks represent different domains of cognitive function: working memory and executive function. Concurrent validity will be studied to validate the dual-task walking measures with each other and with the item 14 of the mini-Balance Evaluation Systems test (Mini-BESTest) and dual-task Timed-up-and-Go test (dual-TUG) obtain concurrently for assessing dual-task ability. In addition, we will compare dual-task walking performance between fallers and non-fallers to examine discriminant validity of dual-task assessments.

A comparative efficacy research is a single-blind, randomized controlled trial. Sixty stroke patients will be randomized to MCDTT or MDTT or CDTT. All three groups will receive dual-task interventions at progressively increasing task difficulty 3 times a week for 4 weeks. The MCDTT group will undertake sitting to standing, standing balance, and treadmill walking training while concurrently perform motor and cognitive tasks. The MDTT and the CDTT groups will train the same set of sitting to standing, standing balance, and walking activities as the MCDTT group while simultaneously performing only motor or cognitive task, respectively. During each session, all participants will receive the instruction of a variable priority to practice shifting attention between tasks by spending half of the training attention focus on the balance task, and half focus on the secondary cognitive or motor tasks. A blinded assessor will administer three assessments All participants will be examined gait and cognitive performance under single-task (walking only, cognitive tasks only) and dual-task conditions (walking while performing 3 cognitive tasks) at two baselines, post intervention, and 1-month follow-up. The primary outcome measure of gait and cognition is gait speed and composite score of accuracy and reaction time of the cognitive tasks under single- and dual-task conditions. The secondary outcome measures will be the Berg Balance Scale, Mini-BESTest, dual-TUG, Functional Gait Assessment, Activity-specific Balance Confidence Scale, Chair Stand Test, Stroke Impact Scale, and Patient Global Impression of Change. Repeated measure ANOVA will be used to compare measurements at baseline, after training, and follow-up among the groups.

Number of Planned Patients: 60 stroke patients Duration of the Study: 2018/08/01～2021/07/31

ELIGIBILITY:
Inclusion Criteria:

* (1) first-ever stroke with onset duration more than 3 months
* (2) able to walk 10 m
* (3) no severe vision, hearing, and language problems.

Exclusion Criteria:

* orthopedic and other neurological disorders that affect walking
* other treatments that could influence the effects of the interventions (e.g., recent Botulin toxin treatment of the lower extremity)
* moderate or severe cognitive impairments (score < 24 on Mini-Mental State Examination)
* severe uncorrected visual deficits.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
gait speed | 10 minutes
  Participants will walk 10m at their preferred speed and at fast speed. A 12-meter walkway will be used for walking testing. In order to allow the subjects to have enough distance to accelerate and decelerate, only the time taken to walk the middle 10 meters will be recorded by a stopwatch. The primary gait parameter is gait speed (cm/s) under dual-task walking conditions using the 10 Meter Walking Test.
composite score | 10 minutes
  For all the cognitive tasks, we will calculate a composite score for cognitive-task performance by dividing the accuracy (% correct responses) with the reaction time of correct answers (milliseconds), which accounts for speed-accuracy tradeoffs in the overall dual-task effect.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS). | 5-10 minutes
  The BBS is a 14-item scale quantitatively assesses both static and dynamic balance with psychometrically sound measure of balance impairment after stroke. The items are scored from 0 to 4, with a score of 0 representing independent item completion. Scores of the BBS range from 0 to 56, with higher scores suggest better balance.
Mini-Balance Evaluation Systems Test (Mini-BESTest). | 10 minutes
  The Mini-BESTest consists of 14 items and.includes four subscales: anticipatory postural adjustmentsl, reactive postural control, sensory orientation, and dynamic gait. Each item is rated on a three-point ordinal scale (0 = severe, 1=moderate, and 2 = normal), with a maximum score of 28 points.
Timed Up and Go Test (TUG) | 2 minutes
  The TUG test will be used as an index of dynamic balance of the elderly and stroke patients. At the signal, participants stand up, walk 3 m, turn, walk back, and sit down again. The score is the time to complete the test measured using a stopwatch. The TUG test will be administered under the single-task (preferred speed and maximum fast) and dual-task conditions (tray carrying and counting backward by 3s). In dual-task condition, participants will be asked to perform the TUG test while carrying a tray with glasses (dual-TUG manual) or counting backward by 3s (dual-TUG cognition). The instruction for dual-TUG tests is to walk with your comfortable speed and concurrently perform a secondary task (carry the tray in front of you with both hands without dropping glasses on the tray or counting backward by 3s).
Functional Gait Assessment (FGA). | 10 minutes
  The FGA is comprised of 10-item that contains 7 of 8 items (except walking around obstacles) from the Dynamic Gait Index and 3 additional tasks, including walking with a narrow base of support, walking with the eyes closed, and walking backward. Subjects' performance of each test item was rated on a 4-point scale (0-3), with the total score ranging between 0 and 30.
Activity-specific Balance Confidence Scale (ABC). | 2 minutes
  The ABC will be used to determine fear of falling and self-reported confidence when performing 15 different daily activities, such as walking around the house, walking up and down stairs, and walking on slippery floors. A confidence rating scale ranges from 0% to 100%, with 0% indicating no confidence, and 100% indicating full confidence.
Chair Stand Test (CS). | 2 minutes
  The Chair Stand Test measures lower extremity muscular strength.87 The participants will be instructed to stand from a seated on the chair position as much as possible for 30 seconds. The total number of stands was counted in 30 seconds. Timed five-chair stand (TCS) is the time measured using a stopwatch to complete five times of standing from sitting
Muscle Strength of Lower-Extremity. | 10 minutes
  Handheld dynamometers (MicroFET2, Hoggan Health Industries Inc, West Jordan, Utah; Jamar ® Plus+ hand dynamometer, Patterson Medical® Sammons Preston®) will be used to measure the maximum isometric strength of tibialis anterior and grip strength (averaged over three attempts and left and right limbs) using a standard protocol with high test-retest reliability.
Patient Global Impression of Change Scale (PGIC). | 1 minutes
  Participants will be evaluated regarding the participants' perception with the change in balance and gait related to the intervention. The PGIC is a transition scale that is a single question asking the patients to rate their balance/gait now, as compared with how it was prior to before beginning treatment on a scale from 1 (very much better ) to 7 (very much worse).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No